CLINICAL TRIAL: NCT00998855
Title: Glucose and Lipid Metabolism in Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institutes of Health (NIH) (NIH)
Responsible Party: Agneta L Sunehag M.D., Ph.D., Baylor College of Medicine, Houston TX
Organization: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: sunehagexercise; NIHNICHDRO1 HD044609
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2009-10

CONDITIONS: Exercise; Obesity; Insulin Sensitivity
Keywords: Exercise in obesity
MeSH Terms: conditions — Motor Activity; Obesity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescents: Post pubertal, sedentary lean and obese Hispanic adolescents
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 12 wk aerobic or/ resistance exercise program

SUMMARY:
A 12 wk aerobic exercise program will reduce visceral, hepatic and intramyocellular fat accumulation and improve insulin sensitivity and glucose metabolism in obese sedentary Hispanic adolescents.

DETAILED DESCRIPTION:
Lean and Obese post pubertal adolescents perform an aerobic exercise program 30 minx4/week at a heart rate corresponding to at least 70% of that obtained at VO2 peak. The exercise program is preceded and followed by a 7 d diet delivered by the metabolic research kitchen (identical on both study occasions); metabolic studies (identical on both study occasions) including 24h calorimetry, measurements of glucose and lipid metabolism and insulin sensitivity and secretion using compounds labelled with stable i.e. non radioactive isotopes and gas chromatography-mass spectrometry.Fat mass and lean body mass are measured by DXA and visceral/subcutaneous, hepatic and intramyocellular fat by MRI/MRS. Since we want to specifically determine the effects of exercise, there is no intent of weight loss. The subjects are weighed twice a week to assure weight stability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No medication
* Sedentary
* No first degree relative with diabetes,
* Hispanic
* BMI >30 or <25 kg/m2.

Exclusion Criteria:

* Any medication including birth control pills
* Performing more than >45 min of moderate to light physical activity/week
* Chronic illness

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Sedentary, post pubertal, Hispanic lean and obese adolescents
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2004-02; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Fat distribution, insulin sensitivity, glucose production, gluconeogenesis, glycogenolysis | In response to a 12 wk exercise program.

SECONDARY OUTCOMES:
Lipolysis, blood lipids, adiponectin, leptin and CRP | In response to a 12 wk exercise program

CONTACTS AND LOCATIONS:
Overall Officials: Agneta L Sunehag, M.D., Ph.D, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States